CLINICAL TRIAL: NCT02621632
Title: SocknLeg - a User Friendly Medical Compression Study of a Modified Application of a Medical Device
Acronym: Socknleg
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: KEK-ZH-Nr. 2013-091
Record Dates: First submitted 2015-05-22; First posted 2015-12-03 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Venous Insufficiency
Keywords: Compression therapy
MeSH Terms: conditions — Venous Insufficiency

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Healthy subjects and patients (Other): To done a novel compression system. 20 healthy subjects and 20 patients done a novel compression system termed Socknleg and a compression class III stocking as a comparator.The Socknleg compression system was developed by the investigator and produced by Sigvaris AG, St. Gallen, Switzerland.
  Interventions: Device: (Socknleg)To done of a novel compression system

INTERVENTIONS:
Device: (Socknleg)To done of a novel compression system — To done a novel compression system.

SUMMARY:
The study intends to investigate a novel compression system termed Socknleg composed of an understocking covering the foot with three added stockings extending from the ankle to the knee without covering the foot. The novel Socknleg system is compared to a standard class III compression stocking.

DETAILED DESCRIPTION:
The investigator tests a novel compression system termed Socknleg in 20 healthy individuals and 20 patients with chronic venous disease. Socknleg is composed of an understocking covering the foot with three added stockings extending from the ankle to the knee without covering the foot. The novel Socknleg system is compared to a standard class III compression stocking. Outcome measures are successful donning and the comparison of interface pressure measured on the level of the ankle.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers: age > 18 years, proband information read, consent form signed
* Patients: age > 18 years, chronic venous insufficiency CEAP C5 (healed venous ulcer).Age > 18 year, patient information read, consent signed.

Exclusion Criteria:

* Active venous ulcer
* Peripheral arterial disease
* Peripheral neuropathy

Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2013-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Donning success. | Successful donning has to be completed within 5 minutes.
  Ability to fully done the investigated compression devices.

SECONDARY OUTCOMES:
Interface pressure | Interface pressure is measured within 5 minutes of complete donning of the stocking.
  Interface pressure of the compression systems is measured at level cB1 (transition of the Achilles tendon to the calf muscle) in mmHg by a pressure measuring device termed Picopress® . Interface pressure is compared between the novel compression system and the comparator, a class III compression stocking.

CONTACTS AND LOCATIONS:
Overall Officials: Juerg Hafner, Prof. (MD), Principal Investigator — University of Zurich
Locations (1):
- Department of Dermatology, University Hospital of Zurich, Switzerland, Zurich, Canton of Zurich, Switzerland